CLINICAL TRIAL: NCT03367962
Title: Detection of Graft Versus Host Disease With [18F]F-AraG, a Positron Emission Tomography Tracer for Activated T Cells
Brief Title: Detection of Graft Versus Host Disease With [18F]F-AraG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: Stanford University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB_38850; 5P01CA049605 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Graft Versus Host Disease
Keywords: PET-CT scan; [18F]F-AraG
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Highly suspected to already have aGVHD (Experimental): Patients highly suspected to have aGVHD. These patients will undergo a [18F]F-AraG PET-CT scan following a biopsy taken to confirm aGVHD.
  Interventions: Drug: [18F]F-Ara-G
- High risk of developing aGVHD (Experimental): Patients at high risk of developing aGVHD will undergo a [18F]F-AraG PET-CT scan on day 4 +/- 2 days post transplant. Additionally these patients will be scanned again between day 14-21 post transplant.
  Interventions: Drug: [18F]F-Ara-G
- Healthy Subjects (Experimental): Healthy subject volunteers will undergo preliminary evaluation to ensure eligibility, receive and sign an informed consent, be enrolled in the trial, and then have a [18F]F-AraG PET-CT scan.
  Interventions: Drug: [18F]F-Ara-G

INTERVENTIONS:
Drug: [18F]F-Ara-G — the [18F]F-AraG tracer will be administered as a single bolus injection of approximately 5 mCi into a hand or arm vein.

SUMMARY:
This is a single-center imaging study to determine utility of in vivo imaging with [18F]F-AraG to identify sites of Graft Versus Host Disease (GVHD) in patients highly suspected of having acute GVHD who require systemic therapy, and patients at high risk for developing acute GVHD. [18F]F-AraG PET scans will be compared to biopsy results to correlate T cell accumulation which is implicated in the disease. High risk patients will be followed to verify predictive potential of [18F]F-AraG.

DETAILED DESCRIPTION:
This single-center imaging study will enroll three cohorts of participants: healthy volunteers, patients highly suspected to have acute GVHD (aGVHD) and requiring systemic therapy, and patients at high risk for developing GVHD.

A total of 5 healthy volunteers will undergo [18F]F-AraG PET scans and blood sampling to better understand [18F]F-AraG biodistribution and stability in the body.

A total of 10 highly suspected acute GVHD patients will be scanned following biopsy taken to confirm aGVHD. The staging and grading of the disease using the Glucksberg grade and International Bone Marrow Transplant Registry Severity Index (IBMTR) at time of enrollment will be noted. Biopsy tissues of consented patients will be analyzed further for T cell involvement.

A total of 15 high-risk patients (recipients of myeloablative or reduced intensity allogeneic transplants using either bone marrow or peripheral blood stem cells from HLA-matched or HLA-mismatched related or unrelated donors-protocols 9142, 9022, 9924) will be recruited. All those that consent will undergo a PET-CT scan with [18F]FAraG on day 4 +/- 2 days post transplant. Additionally, these patients will be scanned again between day 14-21 post transplant. Follow up on these patients will note those that go on to develop aGVHD and the clinical end point will be correlated to the scans to verify the predictive potential of the radiotracer.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 21 years of age or older.
2. Must understand and voluntarily have signed an Informed Consent after its contents have been fully explained.

   1. For patients highly suspected to have aGVHD and requiring systemic therapy, informed consent should be signed after biopsy taken to support clinical diagnosis.
   2. For patients at high risk for developing aGVHD, informed consent should be signed prior to transplant.
3. For healthy volunteers only: Must have no known medical problems that would make undergoing the scan hazardous to the health of the patient or interfere with the results. In particular subjects should not have any cardiac or immunological disorders as these would likely affect the scan results. Subjects should have had a full physical exam within 6 months of the study. If healthy volunteers have not had a full medical exam within 6 months of the study, one of the nuclear medicine physicians will conduct the medical exam prior to any study procedures.
4. For patients highly suspected to have aGVHD and requiring systemic therapy only: Taking steroid treatment for suspected aGVHD for 3 days or less.
5. For patients at high risk for developing aGVHD only: Recipients of myeloablative or reduced intensity allogeneic transplants using either bone marrow or peripheral blood stem cells from HLA-matched or HLA-mismatched related or unrelated donors (protocols 9142, 9022, 9924) who have not yet been placed on any therapy for acute GVHD.

Exclusion Criteria:

1. Pregnant or nursing
2. Individuals with known or suspected substance abuse, obtained by self-reporting.
3. Uncontrolled infection
4. Relapsed/persistent malignancy
5. Currently receiving immunotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Negrin, M.D.., Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Highly Suspected to Already Have aGVHD | High Risk of Developing aGVHD | Healthy Subjects
Started | 7 | 2 | 0
Completed | 6 | 2 | 0
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ran out of funding for Healthy Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Highly Suspected to Already Have aGVHD | High Risk of Developing aGVHD | Healthy Subjects | Total
Number analyzed (Participants) | 7 | 2 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 0 | 9
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5
  Male | 4 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 2 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 1 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Acute GVHD Grades (MAGIC Criteria) at Time of PET/CT Scan
Description: Acute GVHD severity was graded using the Mount Sinai Acute GVHD International Consortium (MAGIC) criteria (Grades I-IV). Grades were assigned based on organ involvement documented in the clinical chart and biopsy review at the time of the PET/CT scan. We reported the number of participants within each grade.
Time Frame: At the time of the PET/CT scan: within 7 days of GVHD suspicion for the Highly Suspected arm, and at the Day 4 ± 2 post-transplant scan for the High-Risk arm
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Suspected to Already Have aGVHD | High Risk of Developing aGVHD
Number analyzed (Participants) | 6 | 2
Participants
  Grade 0 | 0 | 2
  Grade 1 | 0 | 0
  Grade 2 | 4 | 0
  Grade 3 | 1 | 0
  Grade 4 | 1 | 0

2. Primary Outcome: Number of Participants Who Developed aGVHD Within 6 Months Post-Scan.
Description: All participants were followed for 6 months post-imaging. Development of GVHD was defined by clinical diagnosis documented in the medical record..
Time Frame: From PET/CT scan to 6 months post-scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Highly Suspected to Already Have aGVHD | High Risk of Developing aGVHD
Number analyzed (Participants) | 6 | 2
Participants | 6 | 2

3. Secondary Outcome: Biodistribution and Kinetic Behavior of [18F]F-AraG in Healthy Volunteers
Description: This outcome was intended to assess biodistribution and kinetic behavior of [18F]F-AraG in healthy adult volunteers. However, no healthy volunteers were imaged due to funding limitations.
Time Frame: Follow up will occur 2 to 7 days post scan.
Population: No healthy volunteers were imaged due to loss of study funding; therefore, no data were collected for this outcome.
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 7 days after the single tracer infusion in the "Highly Suspected to Already Have aGVHD" Arm and **up to 7 days after the first and final scan in the "High Risk of Developing aGVHD" Arm".
Description: No participants experienced adverse events
Arm/Group | Highly Suspected to Already Have aGVHD | High Risk of Developing aGVHD | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT03367962/Prot_SAP_000.pdf